CLINICAL TRIAL: NCT04872712
Title: Comparison of the Effectiveness of Manual Acupuncture Therapy Between Press Needle and Filiform Needle for Symptoms of Insomnia and Melatonin Hormone Serum on COVID-19 Frontline Health Workers at RSCM.
Brief Title: Comparing Press and Filiform Needle Acupuncture Effectiveness for Improving Insomnia in COVID-19 Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. Irma Nareswari, B.MedSc, Sp.Ak, Head of Medical Acupuncture Study Programme University of Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-02-0142
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Insomnia
Keywords: Acupuncture; Press Needle; Insomnia; Healthcare worker
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator do not know the respondents. There will be 3 Outcomes Assessors who will randomly assess the respondents. The laboratory assistant will not be informed of the treatments provided to the respondents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Press Needles (Active Comparator): The subjects/population of this study is Health Workers with insomnia symptoms who work at at Cipto Mangunkusumo Hospital treating COVID-19 patients. Subjects group with Press Needles treatment will be treated with 2-week needle retention, 20-second pressing 3 times a day and needle replacement performed every 5 days. The needles are inserted 0.9 mm deep at the acupuncture points HT7 Shenmen, PC6 Neiguan, ST36 Zusanli and SP6 Sanyinjiao.
  Interventions: Procedure: Press needles
- Filiform Needles (Active Comparator): The subjects/population of this study is Health Workers with insomnia symptoms who work at at Cipto Mangunkusumo Hospital treating COVID-19 patients. Subjects group with filiform needles treatment will be treated with 20-minute needle retention, 3 times a week for 2 weeks (total of 6 therapy sessions). The needles are inserted approximately 12 mm deep at the acupuncture points HT7 Shenmen and PC6 Neiguan and 25 mm deep at the ST36 Zusanli and SP6 Sanyinjiao.
  Interventions: Procedure: Filiform Needles

INTERVENTIONS:
Procedure: Press needles — Manual acupuncture using press needles
  Arms: Press Needles
Procedure: Filiform Needles — Manual acupuncture using filiform needles
  Arms: Filiform Needles

SUMMARY:
The purpose of this study is to compare the effectiveness of manual acupuncture between 2 types of needles in subsiding insomnia symptoms of healthcare workers who were responsible for treating COVID-19 Patients in Cipto Mangunkusumo hospital.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of manual acupuncture between press needles and filiform needles for subsiding insomnia symptoms based on changes in the Pittsburgh Sleep Quality Index (PSQI) questionnaire score and examination of Melatonin in blood. If the press needles proven to be superior, this method would also be more beneficial during this pandemic as this can shorten the time and/or frequency of the therapy sessions, hence reducing interaction and risk of COVID-19 transmission.

ELIGIBILITY:
Inclusion Criteria:

* Health care workers treating COVID-19 patients in Cipto Mangunkusumo Hospital.
* Has Symptoms of insomnia for at least 2 weeks (screened using the PHQ-9 instrument modified to question number 3a with an answer score of at least 1)
* Age 20 - 50 years.
* Has negative COVID-19 rapid test or PCR swab result in the 7 days prior to the study.
* Willing to participate in research by signing an informed consent.
* Willing to follow the research process to completion.

Exclusion Criteria:

* If you answered Yes to PHQ-9 number 3a never or 3b with a yes
* Insomnia is caused by moderate pain (with Numeric Rating Scale > 4)
* Insomnia patients with medical therapy such as benzodiazepines, non-benzodiazepines, melatonin drugs and antidepressants
* Has severe social and occupational dysfunction (with the Global Assessment of Functioning < 50).
* Has a history of contraindications to acupuncture such as medical emergencies, pregnancy, thrombocytopenia with a platelet count below 50,000 per microliter of blood, history of blood clotting disorders / taking blood thinners, puncturing over malignant tumors, or infection or scarring in the acupuncture area.
* The patient is febrile with a temperature more than 38 Celsius
* Have had acupuncture in the last 7 days prior to study.
* No limbs
* Cognitive impairments or impaired consciousness

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) Questionnaire Score | 6 weeks (4 times measurement : Before the treatment and every 2 weeks until week 6)
  Pittsburgh Sleep Quality Index (PSQI) Questionnaire used have 19 questions related to sleep quality and disturbances, grouped into seven-component scores. The seven components of the score were then summed to produce the global PSQI score, which has a range from 0 as minimum and 21 as maximum score. Higher Total PSQI score indicates poorer sleep quality.
  The PSQI score was measured at 4 time points per subject (Before the treatment and every 2 weeks until week 6) to understand the change and impact before and after the treatment as well as the lasting effect within 4 weeks of treatment was finished.
Change in Melatonin Level via Blood Test | 2 weeks ( 2 times measurement : Before the treatment and after the treatment is completed (treatment duration: 2 weeks)
  Melatonin Level was measured through blood sampling and test to determine the level of melatonin (in pg/mL) in the human serum. The higher the Melatonin Level indicates better outcome.
  The Melatonin Level was measured 2 times for all subjects (Before and after the treatment which is in span of 2 weeks) to understand the change and impact before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Irma Nareswari, dr. Sp.Ak, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No